CLINICAL TRIAL: NCT03632850
Title: Shared Decision-making: Investigating the Potential of an Interactive, Web-Based, Information Tool for People With Advanced Pancreatic Cancer
Brief Title: Web-based Treatment Information Tool for People With Advanced Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Poole Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 252843
Record Dates: First submitted 2018-07-25; First posted 2018-08-16 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Advanced Pancreatic Cancer
Keywords: pancreatic cancer; shared decision-making; decision aids; web-based decision tool; mixed methods
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Doctors: This is a group of oncologists who have experience in treatment deliberations with patients of advanced cancer.
  Interventions: Other: web-based interactive tool
- Nurses: This is a group of clinical nurse specialists who have experience in treatment deliberations with patients of advanced cancer
  Interventions: Other: web-based interactive tool
- Patients: this is a group of adult patients who have been diagnosed with advanced pancreatic cancer
  Interventions: Other: web-based interactive tool
- Relatives: this is a group of adults who are involved in providing support for their loved ones who are diagnosed with advanced pancreatic cancer
  Interventions: Other: web-based interactive tool

INTERVENTIONS:
Other: web-based interactive tool — an online tool to assist users in decision-making in choice of treatment for advanced cancer

SUMMARY:
Pancreatic cancer (PC) is usually diagnosed at a late stage when it is incurable, thereby limiting treatment to palliative care. Chemotherapy is one of the standard palliative care options. Due to the availability of different regimens with varying degrees of benefits and risks, clinicians and patients with advanced pancreatic cancer usually discuss treatment options in order to arrive at the most appropriate chemotherapy regimen for the patient. The use of information tools has produced positive results in explaining the benefits and risks of different treatment options for diseases like stage IV lung cancer, ovarian cancer, and colorectal cancer. However, there is no such tool for people with advanced pancreatic cancer. With over 80% of people with pancreatic cancer being diagnosed in the advanced stage, it would be beneficial to enhance effective decision-making with respect to treatment at this challenging time of the disease progression.

The aim of this research is to investigate the potential of a web-based information tool to support decision-making about treatment options for people who have been diagnosed with advanced pancreatic cancer.

A multiphase mixed methods design has been adopted for this research study. The identified phases are: (1) systematic review and network meta-analysis of reported randomised controlled trials (RCTs) in advanced pancreatic cancer; (2) focus groups/personal interviews with clinicians, and semi-structured interviews with patients and their relatives; (3) web-based information tool development; and (4) pilot test of the developed information tool with clinicians, patients, and relatives of patients

DETAILED DESCRIPTION:
Pancreatic cancer (PC) is a disease with very low 5-year survival rates. Some estimates set this at less than 5%. In the European Union (EU), over 85,000 deaths were projected in 2017, which is a rise of around 8.0% from 2012. PC can be broadly classified as locally resectable, borderline resectable, locally advanced, and metastatic. Treatments include surgery, chemotherapy, radiation therapy, and palliative care. Surgery offers curative treatment, but 80% of patients are diagnosed in the advanced stage (locally advanced or metastatic) and are ineligible. However, systemic therapy (such as chemotherapy) is a palliative option for people with advanced pancreatic cancer (APC). "Best supportive care" (BSC), or "supportive care", is another option which involves symptom management and improving quality of life.

Shared decision-making (SDM) is a process where clinicians and patients make decisions together using the best available evidence. SDM is recognised as a policy priority and ethical imperative by the National Health Service (NHS) and several healthcare regulators in the United Kingdom (UK), respectively. The concept of equipoise is a scenario where there is more than one legitimate choice of treatment for a medical condition. It offers an opportunity to apply SDM in discussing the choice of treatment for people with APC because there is no clear preference of treatment options in terms of benefits and risks for APC. Moreover, a systematic review in 2006 indicated, among other things, that SDM facilitated positive impact on the clinical process and patient outcomes. Encouraging SDM in APC treatment could yield similar results, including the reduction in selecting aggressive treatments that have little or no corresponding economic or personal benefits.

Several tools have been developed to enhance SDM in relation to other medical conditions. Some of these tools are for ovarian cancer, stage IV lung cancer, and colorectal cancer. CONNECT ™ is a computer-based tool that was developed for the general improvement of the doctor-patient communication process. Additionally, a systematic review in 2015 showed that decision tools can improve patients' knowledge and awareness of the treatment options available to them. However, there is very little in literature about the use of evidence-based digital tools in discussing the expected outcomes of treatment for people with APC. Although predictive tools have been developed for PC, there is currently no web-based information tool that can provide clinical evidence on the treatment choices available to people with APC.

However, there is an online decision aid developed for patients with APC in Canada. It has some useful features which can help its users make decisions about their treatment, including information about APC. However, its automation in comparing treatment options is basic, its depth of information necessary for decision-making, and its flexibility could be improved. Its target audience are the patients only. It also assumes that users typically have only 3 options to choose from, although it suggested the possibility of increasing the user options.

It is necessary that patients are fully aware of the benefits and risks associated with any treatment that is being proposed to them. Also, to ensure that clinicians provide the best available evidence-based information in an easily understandable format for the patients, the purpose of this study is to investigate the potential of an interactive, web-based information tool to facilitate the process of shared decision-making between clinicians, and patients and their relatives (or caregivers).

RESEARCH RATIONALE

1. The need for an evidence-based information tool for APC treatment options:

   There is currently no web-based, SDM tool for APC that presents information on available treatment options in a visual, and concise way to patients so that they and their clinicians can make informed choices. Acceptability and reliability are two important factors to be considered when developing such tools.
2. The support for the policy priority for patient-centred care in the UK:

   In the United Kingdom, shared decision-making is viewed as a priority in patient care. However, effective SDM is enhanced through well-informed participants, and that is an objective of the proposed information tool.
3. Enhancing clinicians' communicative skills:

   Communicative skills was identified in healthcare professionals as a requisite for successful SDM. Therefore, the proposed information tool is hoped to enhance clinicians' capacity to communicate available treatment options with their patients by presenting pertinent facts about APC treatment in a concise and user-friendly manner for them.
4. Improving medical cost-effectiveness This tool could also potentially challenge the "more-is-better" attitude (assumption that expensive treatment equals better healthcare) held by the public. Evaluation of some patient decision aids showed improved cost-effectiveness in some medical conditions. Introducing the information tool to APC treatment could potentially yield similar results.

OBJECTIVES Primary objective To investigate the potential of a web-based, interactive, information tool in facilitating shared decision-making in the choice of treatment for people with advanced pancreatic cancer

Second objectives (i) To assess the quality of life, efficacy, and safety of chemotherapy treatments of APC through systematic review and network meta-analysis (NMA) of randomized controlled trials (RCTs).

(ii) To explore the preferences and expectations of clinicians, people with APC, and their relatives, when making decisions about treatment, through focus groups and semi-structured interviews for clinicians, and people with APC (including their relatives), respectively.

(iii) To identify the features necessary for the design of a web-based information tool to facilitate SDM between clinicians and people with APC about choice of treatment.

(iv) To evaluate the effectiveness of the developed information tool in SDM, through a pilot test with clinicians (doctors and nurse specialists), people with APC, and their relatives.

ELIGIBILITY:
Inclusion Criteria:

* Doctors and nurses must have had experience of a minimum of one consultation with a patient with cancer leading to the administration of chemotherapy
* Patients Diagnosed with advanced pancreatic cancer, Able to speak and understand written English, 18 years or older
* Relatives must be involved in, or aware of, the decision of the patients in choice of treatment, should be responsible for the provision of support to the patient, 18 years or older, Able to speak and understand written English

Exclusion Criteria:

* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be recruited from two settings
  1. NHS sites in England
  2. Pancreatic Cancer UK (PCUK) (for patients and relatives)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | up to 2 weeks after using the web-based information tool
  this is a 16-item validated instrument that measures the effectiveness in, and perceptions around decision making, using the decisional conflict construct, which is a state of uncertainty about the course of action to take. Subscales in the instrument are Informed subscale (3 items), Values Clarity subscale (3 items), Support subscale (3 items), and uncertainty subscale (4 items). The individual score is converted to an equivalent 0-100 scale. A total high score (above 37.5) means a high decisional conflict indicating a poor decision-making outcome, while a score below 25 indicates low decisional conflict hence better decision-making outcome. Mean scores and standard deviations will be reported for this measure.

SECONDARY OUTCOMES:
Usability: System Usability Scale (SUS) | up to 2 weeks after using the web-based information tool
  a measure of the usability of the web-based information tool based on adaptions of the System Usability Scale (SUS).
  This is a 10-item scale with 5 responses per item that measures the ease of use of a system. The scoring involves conversion of the responses to a scale of 100. Scores of 68 or above termed as "above average", while those below 68 are "below average". However, normalization will be done to obtain percentile ranking for the group under investigation.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Royal Bournemouth and Christchurch Hospitals, Bournemouth
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - Poole Hospital NHS Foundation Trust, Poole
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent A, Herman J, Schulick R, Hruban RH, Goggins M. Pancreatic cancer. Lancet. 2011 Aug 13;378(9791):607-20. doi: 10.1016/S0140-6736(10)62307-0. Epub 2011 May 26. PMID 21620466
- [Background] Balaban EP, Mangu PB, Khorana AA, Shah MA, Mukherjee S, Crane CH, Javle MM, Eads JR, Allen P, Ko AH, Engebretson A, Herman JM, Strickler JH, Benson AB 3rd, Urba S, Yee NS. Locally Advanced, Unresectable Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Aug 1;34(22):2654-68. doi: 10.1200/JCO.2016.67.5561. Epub 2016 May 31. PMID 27247216
- [Background] Malvezzi M, Carioli G, Bertuccio P, Boffetta P, Levi F, La Vecchia C, Negri E. European cancer mortality predictions for the year 2017, with focus on lung cancer. Ann Oncol. 2017 May 1;28(5):1117-1123. doi: 10.1093/annonc/mdx033. PMID 28327906
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Ducreux M, Cuhna AS, Caramella C, Hollebecque A, Burtin P, Goere D, Seufferlein T, Haustermans K, Van Laethem JL, Conroy T, Arnold D; ESMO Guidelines Committee. Cancer of the pancreas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v56-68. doi: 10.1093/annonc/mdv295. No abstract available. PMID 26314780
- [Background] Taieb J, Pointet AL, Van Laethem JL, Laquente B, Pernot S, Lordick F, Reni M. What treatment in 2017 for inoperable pancreatic cancers? Ann Oncol. 2017 Jul 1;28(7):1473-1483. doi: 10.1093/annonc/mdx174. PMID 28459988
- [Background] Hui D, De La Cruz M, Mori M, Parsons HA, Kwon JH, Torres-Vigil I, Kim SH, Dev R, Hutchins R, Liem C, Kang DH, Bruera E. Concepts and definitions for "supportive care," "best supportive care," "palliative care," and "hospice care" in the published literature, dictionaries, and textbooks. Support Care Cancer. 2013 Mar;21(3):659-85. doi: 10.1007/s00520-012-1564-y. Epub 2012 Aug 31. PMID 22936493
- [Background] Elwyn G, Laitner S, Coulter A, Walker E, Watson P, Thomson R. Implementing shared decision making in the NHS. BMJ. 2010 Oct 14;341:c5146. doi: 10.1136/bmj.c5146. No abstract available. PMID 20947577
- [Background] Coulter A, Edwards A, Entwistle V, Kramer G, Nye A, Thomson R, Walker E. Shared decision making in the UK: Moving towards wider uptake. Z Evid Fortbild Qual Gesundhwes. 2017 Jun;123-124:99-103. doi: 10.1016/j.zefq.2017.05.010. Epub 2017 May 20. PMID 28532629
- [Background] Edwards A, Hood K, Matthews E, Russell D, Russell I, Barker J, Bloor M, Burnard P, Covey J, Pill R, Wilkinson C, Stott N. The effectiveness of one-to-one risk communication interventions in health care: a systematic review. Med Decis Making. 2000 Jul-Sep;20(3):290-7. doi: 10.1177/0272989X0002000305. PMID 10929851
- [Background] Elwyn G, Edwards A, Kinnersley P, Grol R. Shared decision making and the concept of equipoise: the competences of involving patients in healthcare choices. Br J Gen Pract. 2000 Nov;50(460):892-9. PMID 11141876
- [Background] Gravel K, Legare F, Graham ID. Barriers and facilitators to implementing shared decision-making in clinical practice: a systematic review of health professionals' perceptions. Implement Sci. 2006 Aug 9;1:16. doi: 10.1186/1748-5908-1-16. PMID 16899124
- [Background] Oshima Lee E, Emanuel EJ. Shared decision making to improve care and reduce costs. N Engl J Med. 2013 Jan 3;368(1):6-8. doi: 10.1056/NEJMp1209500. No abstract available. PMID 23281971
- [Background] Veroff D, Marr A, Wennberg DE. Enhanced support for shared decision making reduced costs of care for patients with preference-sensitive conditions. Health Aff (Millwood). 2013 Feb;32(2):285-93. doi: 10.1377/hlthaff.2011.0941. PMID 23381521
- [Background] Elwyn G, Rasmussen J, Kinsey K, Firth J, Marrin K, Edwards A, Wood F. On a learning curve for shared decision making: Interviews with clinicians using the knee osteoarthritis Option Grid. J Eval Clin Pract. 2018 Feb;24(1):56-64. doi: 10.1111/jep.12665. Epub 2016 Nov 16. PMID 27860101
- [Background] Agoritsas T, Heen AF, Brandt L, Alonso-Coello P, Kristiansen A, Akl EA, Neumann I, Tikkinen KA, Weijden Tv, Elwyn G, Montori VM, Guyatt GH, Vandvik PO. Decision aids that really promote shared decision making: the pace quickens. BMJ. 2015 Feb 10;350:g7624. doi: 10.1136/bmj.g7624. PMID 25670178
- [Background] Vogel RI, Petzel SV, Cragg J, McClellan M, Chan D, Dickson E, Jacko JA, Sainfort F, Geller MA. Development and pilot of an advance care planning website for women with ovarian cancer: a randomized controlled trial. Gynecol Oncol. 2013 Nov;131(2):430-6. doi: 10.1016/j.ygyno.2013.08.017. Epub 2013 Aug 27. PMID 23988413
- [Background] Leighl NB, Shepherd FA, Zawisza D, Burkes RL, Feld R, Waldron J, Sun A, Payne D, Bezjak A, Tattersall MH. Enhancing treatment decision-making: pilot study of a treatment decision aid in stage IV non-small cell lung cancer. Br J Cancer. 2008 Jun 3;98(11):1769-73. doi: 10.1038/sj.bjc.6604395. Epub 2008 May 27. PMID 18506180
- [Background] Leighl NB, Shepherd HL, Butow PN, Clarke SJ, McJannett M, Beale PJ, Wilcken NR, Moore MJ, Chen EX, Goldstein D, Horvath L, Knox JJ, Krzyzanowska M, Oza AM, Feld R, Hedley D, Xu W, Tattersall MH. Supporting treatment decision making in advanced cancer: a randomized trial of a decision aid for patients with advanced colorectal cancer considering chemotherapy. J Clin Oncol. 2011 May 20;29(15):2077-84. doi: 10.1200/JCO.2010.32.0754. Epub 2011 Apr 11. PMID 21483008
- [Background] Meropol NJ, Egleston BL, Buzaglo JS, Balshem A, Benson AB 3rd, Cegala DJ, Cohen RB, Collins M, Diefenbach MA, Miller SM, Fleisher L, Millard JL, Ross EA, Schulman KA, Silver A, Slater E, Solarino N, Sulmasy DP, Trinastic J, Weinfurt KP. A Web-based communication aid for patients with cancer: the CONNECT Study. Cancer. 2013 Apr 1;119(7):1437-45. doi: 10.1002/cncr.27874. Epub 2013 Jan 18. PMID 23335150
- [Background] Austin CA, Mohottige D, Sudore RL, Smith AK, Hanson LC. Tools to Promote Shared Decision Making in Serious Illness: A Systematic Review. JAMA Intern Med. 2015 Jul;175(7):1213-21. doi: 10.1001/jamainternmed.2015.1679. PMID 25985438
- [Background] Ansari D, Nilsson J, Andersson R, Regner S, Tingstedt B, Andersson B. Artificial neural networks predict survival from pancreatic cancer after radical surgery. Am J Surg. 2013 Jan;205(1):1-7. doi: 10.1016/j.amjsurg.2012.05.032. PMID 23245432
- [Background] Smith BJ, Mezhir JJ. An interactive Bayesian model for prediction of lymph node ratio and survival in pancreatic cancer patients. J Am Med Inform Assoc. 2014 Oct;21(e2):e203-11. doi: 10.1136/amiajnl-2013-002171. Epub 2014 Jan 20. PMID 24444460
- [Background] Walczak S, Velanovich V. An Evaluation of Artificial Neural Networks in Predicting Pancreatic Cancer Survival. J Gastrointest Surg. 2017 Oct;21(10):1606-1612. doi: 10.1007/s11605-017-3518-7. Epub 2017 Aug 3. PMID 28776157
- [Background] Gresham, G. Informed Decision Making for Patients with Advanced Pancreatic Cancer Considering Chemotherapy: Development and Evaluation of a Clinical Decision Aid for Patients. Université d'Ottawa/University of Ottawa, 2013.
- [Background] Geessink NH, Schoon Y, van Herk HC, van Goor H, Olde Rikkert MG. Key elements of optimal treatment decision-making for surgeons and older patients with colorectal or pancreatic cancer: A qualitative study. Patient Educ Couns. 2017 Mar;100(3):473-479. doi: 10.1016/j.pec.2016.10.013. Epub 2016 Oct 17. PMID 28029569
- [Background] Levinson W, Kallewaard M, Bhatia RS, Wolfson D, Shortt S, Kerr EA; Choosing Wisely International Working Group. 'Choosing Wisely': a growing international campaign. BMJ Qual Saf. 2015 Feb;24(2):167-74. doi: 10.1136/bmjqs-2014-003821. Epub 2014 Dec 31. PMID 25552584
- [Background] O'Connor AM, Llewellyn-Thomas HA, Flood AB. Modifying unwarranted variations in health care: shared decision making using patient decision aids. Health Aff (Millwood). 2004;Suppl Variation:VAR63-72. doi: 10.1377/hlthaff.var.63. PMID 15471770

DOCUMENTS (1):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03632850/Prot_000.pdf